CLINICAL TRIAL: NCT03424083
Title: Contribution of Four Pulmonary Function Tests to Diagnosis in Patients With Respiratory Symptoms in the Primary Care.
Brief Title: Contribution of Four Pulmonary Function Tests to Diagnosis in the Primary Care.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Other Study IDs: B076201731685
Record Dates: First submitted 2018-01-24; First posted 2018-02-06 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 cohort: adult patients of both sexes (>18 and <80 years) with no previous diagnosis or follow up by a pulmonologist, send by a general practitioner to the lung function lab

SUMMARY:
Contribution of four pulmonary function tests to diagnosis in patients with respiratory symptoms in the primary care.

DETAILED DESCRIPTION:
Background Pulmonary function tests are routinely used for the diagnosis of respiratory conditions. Few studies have been conducted, assessing the use of the pulmonary function tests and their contribution to the diagnosis in patients with respiratory symptoms. A recent study in 33 chest services from Belgian hospitals have shown that each of the four common pulmonary function tests (spirometry, lung volume, airway resistance and diffusing capacity) contributes significantly to the final diagnosis made by pulmonologists in new patients with respiratory symptoms.

Primary care physicians however treat the majority of patients with respiratory symptoms and often use a symptom-based approach to make a diagnosis (2). Diagnostic spirometry remains largely underused in primary care and is probably mainly performed in the care of patients with asthma and chronic obstructive pulmonary disease (COPD). Drawbacks of home spirometry also include poorly performed tests and incorrect interpretation of the results (3). In addition, primary care physicians have no access to the three other common pulmonary function tests that contribute independently to the diagnosis of respiratory diseases (1).

Since 2015, our chest service localized in the center of Brussels offers a direct and open access to the lung function laboratory to all the patients referred by their general practitioners. The four common tests are performed in their patients with respiratory symptoms but no clear diagnosis and the patients are not evaluated by the chest physicians. A protocol is however performed with potential advice for additional diagnostic tests (provocation tests, exhaled NO measurement, ergospirometry, imaging,…).

In the present study, we will assess the contribution of the four common pulmonary function tests to diagnosis in patients with respiratory symptoms in the primary care.

Methods Prospective single center cohort study. Adult patients, aged more than 18 years, presenting to the general practitioner with respiratory symptoms but without a clear diagnosis and referred by them for pulmonary function tests will be enrolled in the study. Patients will be excluded if they had diagnosed respiratory disease at our institution and if they are not able to perform pulmonary function testing.

The patients will not be seen or examined by a pulmonologist of the chest service. They will return to the referring family physician for further treatment.

Before lung function testing, the patients will be asked to fill in a questionnaire, including short questions about their medical history and respiratory medications, previous referrals to a pulmonologist, symptoms and comorbidities.

All patients, regardless of the suspected respiratory condition, will also be asked to complete the COPD assessment test (CAT test) to better quantify their symptoms.

The tests (spirometry, plethysmography, airway resistance measurement, diffusion capacity measurement) will then be performed by a qualified lung function lab technician. Interpretation of the results will be made by a pulmonologist. The protocol will be given to the patient or sent to the referring family physician and may also include proposals for additional diagnostic tests.

In second time, one month later, the general practitioner will be contacted by one of the investigators to receive more information about the final diagnosis based on all the investigations done and treatment.

The collected data will be processed in a database and analyzed anonymously. The primary outcome will be the increase in the proportion of diagnosis afforded by the four tests in comparison with spirometry alone. Secondary outcomes will be the proportion of patients without clear diagnosis, time to lung function tests and time to diagnosis.

Statistical analysis The present study is mainly descriptive and no hypothesis can be made on the contribution of additional lung function tests to the final diagnosis in a population of patients from general practitioners. The present study will include 100 patients with respiratory symptoms but no clear diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* all subjects: 18 or older than 18 years old and younger than 80 years old
* send by a general practitioner for a lung function test

Exclusion Criteria:

* subjects, younger than 18 years old
* not able to perform the lung function tests
* incomplete lung function tests
* disease already diagnosed
* already follow up by a pulmonologist
* preoperative test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * all patients, send by a general practitioner to our lung function lab
  * adults patients (older than 18 years and younger than 80 years), both sexes
  * not followed by a pulmonologist
  * no previous diagnosis and established treatment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-07-25 (Estimated); Study Completion 2018-09-25 (Estimated)

PRIMARY OUTCOMES:
number of cases in which the four lung function tests are contributing to the final diagnosis | at study completion
  number of cases in which the four lung function tests are contributing to the final established diagnosis compared to spirometry alone

SECONDARY OUTCOMES:
number of cases in which additional tests were performed | at study completion
  number of cases in which additional tests were needed to establish the correct final diagnosis, after the performance of the four lung function tests
changes in treatment after the four lung function tests | at study completion
  changes in treatment, prescribed by the primary physician, after the performance of the four lung function tests

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ninane, M.D., PhD, Principal Investigator — CHU St Pierre
Locations (1):
- CHU St Pierre, Brussels, Belgium